CLINICAL TRIAL: NCT02691481
Title: Effect of Diabetes-specific Formulas on Glucose Metabolism and GLP-1 Secretion in Patients With Type 2 Diabetes
Brief Title: Diabetes-Specific Nutritional Formulas Versus Oatmeal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2014-01
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oatmeal breakfast (Active Comparator): consuming 200 kcal of plain cooked oatmeal for breakfast
  Interventions: Dietary Supplement: Oatmeal breakfast; Dietary Supplement: Glucerna formula; Dietary Supplement: Ultra Glucose Control formula
- Glucerna formula (Active Comparator): consuming 200 kcal of Glucerna shake for breakfast
  Interventions: Dietary Supplement: Oatmeal breakfast; Dietary Supplement: Glucerna formula; Dietary Supplement: Ultra Glucose Control formula
- Ultra Glucose Control formula (Active Comparator): consuming 200 kcal of Ultra Glucose Control shake for breakfast
  Interventions: Dietary Supplement: Oatmeal breakfast; Dietary Supplement: Glucerna formula; Dietary Supplement: Ultra Glucose Control formula

INTERVENTIONS:
Dietary Supplement: Oatmeal breakfast
Dietary Supplement: Glucerna formula
Dietary Supplement: Ultra Glucose Control formula

SUMMARY:
Diabetes-specific nutritional formulas (DSNFs) are frequently used as part of medical nutrition therapy for patients with type 2 diabetes in order to improve glycemic control and enhance weight reduction. The mechanism through which DSNFs improve postprandial (PP) plasma glucose is not yet known.

The aim of this study is to compare the effects of 2 DSNFs versus oatmeal on PP plasma glucose, serum insulin and serum active glucagon-like peptide-1 (GLP-1), serum free fatty acids (FFA) and serum triglycerides (TG).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes treated with oral diabetes medications

Exclusion Criteria:

* Type 1 diabetes

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve 0-240 minutes | 240 minutes

IPD SHARING:
Plan to Share IPD: No